CLINICAL TRIAL: NCT03973086
Title: A Double-blind, Randomized, Placebo-controlled Study to Assess the Efficacy of CitruSlim® on Body Composition as Well as Metabolic and Hormonal Factors in Overweight and Obese Individuals
Brief Title: To Assess the Efficacy of CitruSlim® on Body Composition as Well as Metabolic and Hormonal Factors in Overweight and Obese Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HP/190201/CITRUSLIM/BCMH
Record Dates: First submitted 2019-05-07; First posted 2019-06-04 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2019-06

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Citrus flavonone-O-glycosides (Low dose) (Experimental)
  Interventions: Dietary Supplement: Citrus flavonone-O-glycosides- LD
- Citrus flavonone-O-glycosides (High dose) (Experimental)
  Interventions: Dietary Supplement: Citrus flavonone-O-glycosides- HD
- Microcrystaline Cellulose- 400mg (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Citrus flavonone-O-glycosides- LD — Low Dose of 200 mg
  Arms: Citrus flavonone-O-glycosides (Low dose)
Dietary Supplement: Citrus flavonone-O-glycosides- HD — High Dose of 400 mg
  Arms: Citrus flavonone-O-glycosides (High dose)
Dietary Supplement: Placebo — Placebo (Microcrystalline Cellulose) of 400 mg
  Arms: Microcrystaline Cellulose- 400mg

SUMMARY:
CitruSlim® can promote healthy weight loss by promoting anabolic state during weight loss programs, prevent the body from storing fat, reduce appetites and maintain healthy cholesterol and blood glucose level during weight loss program.

This study focuses to prove the efficacy and safety of the product in a population of overweight and obese individual.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants with the age of ≥18 and ≤ 60 years of age.
2. BMI of ≥25 - ≤ 35 kg/m2
3. Waist circumference:India: Men: > 94 cm (37 inches), Women: >80 cm (31.5 inches) USA: Men: > 102 cm (40 inches), Women: >89 cm (35 inches)
4. Triglycerides >150 mg/dL
5. Blood pressure: Systolic: ≥130 mm Hg and/or Diastolic: ≥85 mm Hg
6. Fasting blood glucose ≥ 100 mg/ dl
7. Low HDL level: Men: < 40 mg/dL, Women: < 50 mg/dL
8. Ready to give voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

Participants meeting any of the following criteria will be excluded from the trial:

1. Current smoker.
2. Inability to walk independently.
3. Presence of unstable, acutely symptomatic, or life-limiting illness.
4. Neurological conditions causing functional or cognitive impairments
5. Unwillingness or inability to be randomized to one of three intervention groups.
6. Bilateral hip replacements.
7. Exposure to any non-registered drug product within 3 months prior to the screening visit.
8. Unable/unwillingness to complete study specific diaries (digital/paper-based).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
Change in body fat percent Body Mass Index (kg/m2) | 16 weeks.
  Assessed using DEXA
Change in Lean Body Mass (g) | 16 weeks
  Assessed using DEXA
Change in Body Fat (%) | 16 weeks
  Assessed using DEXA
Change in Fat Free Mass (g) | 16 weeks
  Assessed using DEXA

CONTACTS AND LOCATIONS:
Locations (1):
- Reveal, Bradenton, Florida, United States

IPD SHARING:
Plan to Share IPD: No